CLINICAL TRIAL: NCT00491738
Title: A Multicenter, Phase II, Randomized, Blinded, Placebo-Controlled Trial Evaluating the Efficacy and Safety of Sutent With or Without Bevacizumab in First-Line Patients With Metastatic Renal Cell Cancer
Brief Title: A Study Evaluating the Efficacy and Safety of Sunitinib With or Without Bevacizumab in First-Line Patients With Metastatic Renal Cell Cancer (SABRE-R)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on the data collected, the combination of bevacizumab and sunitinib appeared to be poorly tolerated.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Frank A. Scappaticci, M.D., Ph.D., Study Director, Genentech, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVF4167g
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Results first posted 2009-04-10 (Estimated); Last update posted 2009-04-10 (Estimated); Status verified 2009-04

CONDITIONS: Renal Cell Carcinoma
Keywords: RCC; Renal cell cancer; Avastin; Sutent
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Bevacizumab; Sunitinib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: bevacizumab; Drug: sunitinib
- 2 (Placebo Comparator)
  Interventions: Drug: sunitinib; Drug: placebo

INTERVENTIONS:
Drug: bevacizumab — Intravenous repeating dose
  Arms: 1
Drug: sunitinib — Oral repeating dose
Drug: placebo — Intravenous repeating dose
  Arms: 2

SUMMARY:
This is a Phase II, multicenter, randomized, blinded, placebo-controlled study designed to evaluate the safety and efficacy of combining bevacizumab with sunitinib relative to placebo with sunitinib in patients with metastatic RCC who have not received prior systemic therapy for metastatic disease. The study will enroll approximately 100 patients at approximately 20 centers in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Histologically confirmed metastatic RCC
* Measurable disease, as defined by RECIST
* Age ≥ 18 years
* ECOG performance status of 0 or 1
* Prior nephrectomy
* Ability and capacity to comply with study and follow-up procedures

Exclusion Criteria:

* RCC with predominantly sarcomatoid features
* Prior systemic or adjuvant therapy for RCC
* Radiotherapy for RCC within 28 days prior to Day 1
* Prior treatment with bevacizumab, sunitinib, sorafenib, axitinib, thalidomide, or other similar agents
* Current need for dialysis
* Life expectancy of < 12 weeks
* Current, recent, or planned participation in an experimental drug study
* Inadequate organ function
* Active infection or fever > 38.5°C within 3 days of starting treatment
* History of other malignancies within 5 years prior to Day 1
* Any other medical conditions (including mental illness or substance abuse) deemed by the clinician to be likely to interfere with a patient's ability to provide informed consent, cooperate, or participate in the study, or to interfere with the interpretation of the results
* Inadequately controlled hypertension
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Class II or greater CHF
* History of myocardial infarction or unstable angina within 6 months prior to Day 1
* History of stroke or transient ischemic attack within 6 months prior to Day 1
* Known CNS disease except for treated brain metastasis
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection) or recent peripheral arterial thrombosis within 6 months prior to Day 1
* History of hemoptysis (≥ 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure or anticipation of need for major surgical procedure during the course of the study
* Serious, non-healing wound; active ulcer; or untreated bone fracture
* Known hypersensitivity to any component of bevacizumab
* Pregnancy (positive pregnancy test) or lactation
* Current, ongoing treatment with full-dose warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-08; Primary Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Scappaticci, M.D., Ph.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + Sunitinib: Intravenous infusion of bevacizumab every 2 weeks at a dose of 10 mg/kg + sunitinib 50 mg/day for 4 weeks, followed by 2 weeks of rest
- Placebo + Sunitinib: Intravenous infusion of placebo every 2 weeks at a dose of 10 mg/kg + sunitinib 50 mg/day for 4 weeks, followed by 2 weeks of rest
Period: Overall Study
Arm/Group | Bevacizumab + Sunitinib | Placebo + Sunitinib
Started | 7 | 9
Completed | 7 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab + Sunitinib | Placebo + Sunitinib | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 7 | 11
  >=65 years | 3 | 2 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 60.4 (11.8) | 58.7 (7.0) | 59.4 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: All Adverse Events (Lab Toxicities Reported Were Only Grade 3 and Higher)
Description: Grades according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v3.0, laboratory toxicities based on local laboratory assessments.
Time Frame: 5 months
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Sunitinib | Placebo + Sunitinib
Number analyzed (Participants) | 7 | 9
participants
  Haemolysis | 1 | 0
  Thrombocytopenia | 1 | 0
  Bradycardia | 1 | 0
  Ear Pain | 1 | 0
  Hypothyroidism | 1 | 0
  Diarrhoea | 3 | 4
  Nausea | 4 | 2
  Vomiting | 1 | 0
  Gastroesphagael Reflux Disease | 2 | 0
  Constipation | 1 | 0
  Dyspepsia | 0 | 1
  Abdominal Distension | 0 | 1
  Stomach Discomfort | 0 | 1
  Oral Pain | 1 | 0
  Fatigue | 3 | 4
  Mucosal Inflammation | 2 | 2
  Pyrexia | 1 | 0
  Infuenza Like Illness | 1 | 0
  Chest Pain | 1 | 0
  Abdominal Abscess | 0 | 1
  Otitis Media | 1 | 0
  Fungal Infection | 1 | 0
  Influenza | 1 | 0
  Sinusitis | 1 | 0
  Contusion | 1 | 0
  Protein Urine | 1 | 0
  Blood Pressure Increased | 0 | 1
  Decreased Appetite | 1 | 0
  Hypoglycaemia | 0 | 1
  Back Pain | 1 | 0
  Musculoskeletal Pain | 1 | 0
  Neck Pain | 0 | 1
  Pain in Extremity | 0 | 1
  Headache | 1 | 3
  Dysgeusia | 1 | 2
  Hypogeusia | 1 | 0
  Dizziness | 0 | 2
  Tremor | 1 | 0
  Anxiety | 1 | 1
  Affect Lability | 1 | 0
  Chromaturia | 0 | 2
  Haematuria | 1 | 0
  Pharyngolaryngeal Pain | 1 | 0
  Throat Tightness | 1 | 0
  Epistaxis | 1 | 0
  Pulmonary Embolism | 1 | 0
  Rash | 4 | 1
  Palmar-Plantar Erythrodysaesthesia | 1 | 2
  Yellow Skin | 2 | 0
  Dry Skin | 1 | 0
  Alopecia | 0 | 1
  Night Sweats | 0 | 1
  Nail Discolouration | 0 | 1
  Petechiae | 1 | 0
  Decubitus Ulcer | 0 | 1
  Urticaria | 1 | 0
  Hypertension | 2 | 3
  Hypertensive Crisis | 1 | 0

LIMITATIONS AND CAVEATS:
Based on the early safety results from this study, Genentech terminated further recruitment and discontinued treatment. Insufficient efficacy information was available to perform additional outcome analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other